CLINICAL TRIAL: NCT02473380
Title: Fluorescence Spectroscopy Guided Surgery for Brain Tumors Resection: a Feasibility Study in Human
Brief Title: Fluorescence Spectroscopy Guided Surgery
Acronym: GLIOSPECT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL14-0270
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Glioma (LGG); High Grade Glioma (HGG)
Keywords: glioma; fluorescence spectroscopy
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraoperative fluorescence spectroscopy (Experimental): The experimental device will be assessed during an open surgical approach for surgical removal of the tumors
  Interventions: Device: Fluorescence spectroscopy guided surgery

INTERVENTIONS:
Device: Fluorescence spectroscopy guided surgery — A prototype of intraoperative fluorescence spectroscope will be used for fluorescence spectroscopy during a surgical procedure (open surgical approach only). The experimental probe dedicated to the spectroscopic system will be positioned against the surface of the brain, emission spectrum will be acquired and measured, and finally compared with anatomopathology exams. One specific medication will be used as contrast agent in the study: 5 amino-levulinic hydrochloride (GLIOLAN, MEDAC) orally at the dose of 20mg/kg of body weight.

SUMMARY:
Intraoperative surgical fluorescence microscopy is a useful technique for the surgical resection of glioma. However the accuracy of this method is limited by its too low sensitivity. Fluorescence spectroscopy has the potential capacity to overcome the current limitations of conventional fluorescence guided surgery by increasing the sensitivity: in a pilot study on brain tumor biopsies, fluorescence spectroscopy was shown to measure two-peaked 5-ALA-induced protoporphyrin IX (PpIX) fluorescence emission spectrum which clearly enables to distinguish the solid component of glioblastomas from low grade gliomas and infiltrative component of glioblastomas. This innovative method could become in future a useful tool for real-time diagnosis of brain lesions (initial diagnosis or follow-up post resection to check for residual dysplasia) and real-time assessment of resections margins during surgery. However, those preliminary ex-vivo results have to be confirmed in a feasibility in-vivo study on human.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Clinical signs and history of the disease in favor of a HGG, LGG
* MRI study in favor of a HGG, LGG, meningioma or brain metastasis
* Affiliated to or beneficiary of a social security system (or equivalent).
* Patients who have provided written informed consent for the study

Exclusion Criteria:

* Previous life-threatening allergic reactions and known hypersensitivity
* Pregnant or lactating or not using effective contraception;
* Restricted renal function define by a creatinine clearance < 30ml/min
* Patients under a beta-blockers treatment
* Contraindication to do an MRI (pace-maker)
* Contraindication to the use of 5-ALA : known hypersensibility to 5-ALA or to porphyrin, acute or chronic porphyria
* Minor or adult ward of court (under guardianship or trusteeship)
* No affiliation to a social security system (or equivalent).
* Patients who express opposition to participation in the study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the feasibility by calculating the ratio of normalized fluorescence intensity measured at 620 nm and at 634 nm | 1 day (End of the surgical procedure)
  The technical feasibility will be assessed by the capacity of the prototype to provide distinguished fluorescence emission spectrum depending on the tumor component (correlation between the spectrum and classical histology).

SECONDARY OUTCOMES:
Assessment of the safety as a composite outcome measure : number, type and severity of recorded adverse events | 14 days after inclusion
  Safety will be assessed by the number, type and severity of recorded adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques GUYOTAT, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Alston L, Mahieu-Williame L, Hebert M, Kantapareddy P, Meyronet D, Rousseau D, Guyotat J, Montcel B. Spectral complexity of 5-ALA induced PpIX fluorescence in guided surgery: a clinical study towards the discrimination of healthy tissue and margin boundaries in high and low grade gliomas. Biomed Opt Express. 2019 Apr 18;10(5):2478-2492. doi: 10.1364/BOE.10.002478. eCollection 2019 May 1. PMID 31149380
- See also: Stummer et al. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol 2006 May;7(5):392-401 — http://www.ncbi.nlm.nih.gov/pubmed/16648043
- See also: Jacquesson et al. [Surgery of high-grade gliomas guided by fluorescence: a retrospective study of 22 patients]. Neurochirurgie. 2013 Feb;59(1):9-16. — http://www.ncbi.nlm.nih.gov/pubmed/?term=23318102
- See also: Montcel et al. Two-peaked 5-ALA-induced PpIX fluorescence emission spectrum distinguishes glioblastomas from low grade gliomas and infiltrative component of glioblastomas. Biomed Opt Express. 2013 Apr 1;4(4):548-58 — http://www.ncbi.nlm.nih.gov/pubmed/23577290